CLINICAL TRIAL: NCT04870151
Title: Anterolateral Versus Direct Lateral Approach in Hemiarthroplasty for Hip Fracture: A Randomised Study
Brief Title: Anterolateral Versus Direct Lateral Approach in Hemiarthroplasty for Hip Fracture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 224045
Record Dates: First submitted 2021-04-19; First posted 2021-05-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hip Fractures
Keywords: Surgical approach; Hemiarthroplasty
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are instructed to assess the outcomes before they log in to the patients' journal. Thereby, they will not have information of the treatment allocation at the time of outcomes assessment. Also, they will not ask the patients to undress or in any other way examine the surgical site, as the location of the scar tissue may disclose the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterolateral approach (Experimental): The minimally invasive anterolateral approach (Watson-Jones approach) is performed with the patient in supine position. An oblique incision is made from just dorsal to the anterior superior iliac spine, and extended distally to the greater trochanter. After the fascia is incised, deep dissection continues in the plane between the tensor fasciae latae and the gluteus medius muscles. The joint capsule is exposed and opened. The femoral head and neck are resected and the femoral canal is reamed according to the preoperative plan.
  A femoral stem (Link Lubinus SPII) is fixed using bone cement (Heraeus Medical Palacos R+G pro) and connected to a bipolar femoral head (Zimmer Multipolar).
  After implantation of the prosthesis, the fascia, subcutis and skin is closed in separate layers with sutures.
  Interventions: Procedure: Anterolateral approach
- Direct lateral approach (Active Comparator): The direct lateral approach (Hardinge approach) is performed with the patient in a lateral decubitus position. A straight or curved longitudinal incision is made over the greater trochanter, and the fascia is incised longitudinally. The anterior aspect of the gluteus medius and minimus muscles are separated from the greater trochanter. The joint capsule is exposed and opened. The femoral head and neck are resected and the femoral canal is reamed according to the preoperative plan.
  A femoral stem (Link Lubinus SPII) is fixed using bone cement (Heraeus Medical Palacos R+G pro) and connected to a bipolar femoral head (Zimmer Multipolar).
  After implantation of the prosthesis, the gluteus medius and minimus muscles are reinserted using osteosutures. The fascia, subcutis and skin is closed in separate layers with sutures.
  Interventions: Procedure: Direct lateral approach

INTERVENTIONS:
Procedure: Anterolateral approach — Cemented hemiarthroplasty using an anterolateral approach.
  Arms: Anterolateral approach
Procedure: Direct lateral approach — Cemented hemiarthroplasty using a direct lateral approach.
  Arms: Direct lateral approach

SUMMARY:
Patients with dislocated hip fractures are randomised to cemented hemiarthroplasty with an anterolateral approach or a direct lateral approach.

DETAILED DESCRIPTION:
Dislocated intracapsular hip fractures are usually treated with cemented hemiarthroplasty. In Norway, a direct lateral approach is most often used, as recommended in national guidelines. In total hip arthroplasty, however, minimally invasive approaches are also commonly used, and may improve the clinical results, as compared to posterior or direct lateral approaches.

The aims of the present study are to evaluate the effect of the minimally invasive anterolateral approach (Watson-Jones approach) compared to the direct lateral approach (Hardinge approach) to the hip joint in hemiarthroplasty after dislocated hip fractures.

Patients with dislocated hip fractures who are fit for cemented hemiarthroplasty are randomised to surgery with an anterolateral approach or a direct lateral approach.

ELIGIBILITY:
Inclusion Criteria:

* dislocated hip fracture.
* planned cemented hemiarthroplasty.
* able to walk, with or without walking aids, prior to the injury.

Exclusion Criteria:

* young and healthy patients with displaced hip fractures who are recommended total hip arthroplasty or open reduction / internal fixation of the fracture.
* patients with severe comorbidity and high risk of cement-related complications who are recommended uncemented hemiarthroplasty (some, but not all, patients with ASA (American Society of Anesthesiologists) grade 4).
* not able to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | 12 months
  Harris Hip Score (HHS) is an outcome measure for hip-related symptoms. The score is based on both patient-reported information and clinical examination, and is administered by a qualified health care professional. It covers four domains: Pain, function, absence of deformity and range of motion. The score ranges from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
EuroQol questionnaire (EQ-5D) | 12 months
  Quality of life is measured by the EuroQol questionnaire (EQ-5D). EQ-5D is a validated generic health-related quality-of-life instrument. It consists of two parts: EQ-5D descriptive part and EQ-5D visual analogue scale. The descriptive part includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with three possible answers ("no problems", "some problems", and "major problems"). EQ-5D VAS is a visual analogue scale of self-related overall health, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Patient-reported limping | 12 months
  Patient-reported limping is a sub-score of the Harris Hip Score. The patients describe their limping as (1) "none", (2) "slight", (3) "moderate" or (4) "severe or unable to walk".
Patient-reported use of walking aid | 12 months
  Patient-reported use of walking aid is a sub-score of the Harris Hip Score. The patients describe their use of walking aid as (1) "none", (2) "cane/walking stick for long walks", (3) "cane/walking stick most of the time", (4) "one crutch", (5) "two canes/walking sticks" or (6) "two crutches or unable to walk".
Trendelenburg test | 12 months
  Trendelenburg test is a clinical test for the integrity of hip abductor muscle function. The test is positive when the patient is unable to maintain the pelvis horizontal to the floor when standing on one leg.
Timed Up and Go (TUG) | 12 months
  The Timed Up and Go (TUG) test is a performance-based measure of functional mobility that was initially developed to identify mobility and balance impairments in older adults.
  The patients start in a seated position, walk 3 meters, turn around, walk back to the chair and sit down. The time starts when the patient is commanded to start and stops when the patient is seated.
Blood loss | During surgery
  The peroperative amount of blood loss (milliliters) is registered
Duration of surgery | During surgery
  The duration of the surgical procedure (minutes) is registered
Length of hospital stay | 12 months
  The length of hospital stay (days) is registered
Adverse events | 12 months
  Adverse events such as perioperative complications, infections, dislocations and reoperations are registered
Mortality | 12 months
  In patients who die within 12 months follow-up, the time of death is registered
Cause of death | 12 months
  In patients who die within 12 months follow-up, the cause of death is registered

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Furunes, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Gjøvik, Innlandet, Norway

IPD SHARING:
Plan to Share IPD: No
We have planned to use all the IPD only within the present study group.